CLINICAL TRIAL: NCT05871736
Title: Cross-cultural Adaptation, Validation and Reliability of Turkish Version of Child Engagement in Daily Life Measure V2 for Children With Cerebral Palsy.
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Hayriye Şimşek, Doctor, Ankara City Hospital Bilkent
Other Study IDs: AnkaraCHBilkentHayriyesimsek01
Record Dates: First submitted 2023-05-10; First posted 2023-05-23 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; participation; self-care; measurement; validity; reliability; cultural adaptation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parents of children with cerebral palsy: Parents of children with CP 1.5-11 years of age who applied to the Physical Medicine and Rehabilitation Clinic of Ankara City Hospital
  Interventions: Other: Turkish version of Child Engagement in Daily Life Measure V2
- Parents of children without cerebral palsy: Parents of healthy children without cerebral palsy 1.5-11 years of age who applied to the Physical Medicine and Rehabilitation Clinic of Ankara City Hospital
  Interventions: Other: Turkish version of Child Engagement in Daily Life Measure V2

INTERVENTIONS:
Other: Turkish version of Child Engagement in Daily Life Measure V2 — Child Engagement in Daily Life Measure V2 will be performed on both groups and GMFCS and MACS levels of children with cerebral palsy will be recorded.

SUMMARY:
Participation in daily activities provides many opportunities for children to improve cognitive, physical and communication abilities. Children's participation in recreational and community activities and performance of self-care activities are considered key processes and outcomes for pediatric rehabilitation. Cerebral palsy (CP), which is one of the most common causes of disability in childhood, is more common in our country than in developed countries. Standardized functional assessment scales should be used to objectively measure participation in daily life activities in children with disability such as cerebral palsy.

The aim of this study is to cross-culturally adapt the the Child Engagement in Daily Life Measure V2 (CEDL) to Turkish language and culture and to examine the structural validity and reliability of the Child Engagement in Daily Life Measure V2 (CEDL) in Turkish children with cerebral palsy.

DETAILED DESCRIPTION:
Purpose:

The aim of this study is to cross-culturally adapt the the Child Engagement in Daily Life Measure V2 (CEDL) to Turkish language and culture and to examine the structural validity and reliability of the Child Engagement in Daily Life Measure V2 (CEDL) in Turkish children with cerebral palsy.

Methods:

Translation and cross-cultural adaptation:

In the present study, permission for the translation and validation process of the CEDL V2 was obtained from the CEDL team at Drexel University. Based on previous studies and guidelines forward and backward translation methods were used to perform the crosscultural adaptation. In Stage 1, two independent professionals translated the CEDL V2 from English to Turkish. After the translated versions were harmonized as a first version (Stage 2) with discussion and consensus of translators and second author, a different bilingual translator with English as her native language performed a backtranslation (Stage 3), who was unfamiliar with and blinded to the original version of the CEDL V2 and the back-translation was reviewed by the developers of the CEDL V2 (Stage 4). In Stage 5, an expert committee, including first and second author, reviewed the prefinal Turkish version of the CEDL V2. Lastly, the prefinal version of the questionnaire was piloted in parents of children with disabilities (n = 30) and without disabilities (n = 30) to determine the clarity of all items and their compatibility for Turkish parents (Stage 6). The Turkish version of the CEDL V2 was finalized as the parents recruited for the pilot study indicated that clarity and understandability of the items were acceptable.

Research design:

A cross-sectional and a single-centre study with a test-retest method and comparison group (children without disability) was conducted to determine the reliability and validity of the Turkish version of the CEDL V2.

Participants:

The study protocol was approved by the Medical Faculty of Yıldırım Beyazıd University Ethics Committee (26379996/28). Based on the principles stated in the Declaration of Helsinki, all subjects were informed about the study and the inform consent was taken from the families.

Parents of children with CP 1.5-11 years of age who applied to the Physical Medicine and Rehabilitation Clinic of Ankara City Hospital will be included in the study. Parents of children with and without CP will be asked to complete the Turkish version of the CEDL V2 if they met the including criteria. Before completing the questionnaires, the sociodemographic characteristics of the parents of children with CP and without CP such as name, surname, age, gender, parent relationship to the child, parent's age, parent's education level, parent's work status, family income (monthly) will be recorded in medical records. Therapists will determine the child's GMFCS ve MACS level through observation and interview with the parent. The participants will be asked to participate in the test-retest component of the study and if they want they will complete the instrument after 2 weeks again. The parents of the children without CP will be asked to complete the measure independently of the primary study participants.

Statistical Analysis The internal consistency of the CEDL scale will be determined by calculating Cronbach's alpha. Rasch analysis will be done by calculating the validity of the questionnaire (construct validity-known groups method) as in the original article. A sample size of 250 patients for Rasch analysis would be able to estimate item difficulty within the range of α=0.05 to ±0.32 logit. This sample size is also sufficient to test for item function difference. A difference of 0.32 between residuals with α=0.05 and β=0.20 Type I and II error values can be detected for any 2 groups .

Latest status:

The study was started on 01.10.2021 at Ankara Bilkent City Hospital , department of Physical Therapy and Rehabilitation in Turkey after approval for the present study had been obtained by the local ethics committee of the Yıldırım Beyazıt University and after the translation and cross-cultural adaptation of the measure had been completed . The measure was filled by parents of 273 children with cerebral palsy and 100 children without cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study,
* They are the parents or caregivers of children
* Their child has a clinical diagnosis cerebral palsy or has no clinical diagnosis
* Their child is 1.5-11 years old during the study
* The person who answered the questionnaire has Turkish literacy

Exclusion Criteria:

* History of orthopedic surgery in the last three months
* Illiterate participants

Ages: 18 Months to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Parents of children with cerebral palsy and children without cerebral palsy 1.5-11 years of age who applied to the Physical Medicine and Rehabilitation Clinic of Ankara Bilkent City Hospital will be included in the study.
Sampling Method: Probability Sample
Enrollment: 373 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Child Engagement in Daily Life Measure V2 | baseline
  Child engagement in daily life measure Version 2( CEDL V2 ) is a 29-item parent proxy-report questionnaire. The questionnaire consists of two domains: (1) Participation in Family and Recreational Activities (Family Rec, 11 items), and (2) Performance of Self-care Activities (Self-care, 18 items) and takes approximately 15 min to complete.
  Two dimensions of Family Rec are rated on a 5-point Likert scale: frequency of participation (5¼very often to 1¼never) and enjoyment of participation (5¼a great deal to 1¼not at all). ,
  Performance of Self-care Activities are rated on a 5-point Likert scale.
  On the scale , higher scores mean a better outcome.
  parents of children with cerebral palsy and parents of children without cerebral palsy will complete the measure at the first data collection point
Child Engagement in Daily Life Measure V2 | two weeks
  Child engagement in daily life measure Version 2( CEDL V2 ) is a 29-item parent proxy-report questionnaire. The questionnaire consists of two domains: (1) Participation in Family and Recreational Activities (Family Rec, 11 items), and (2) Performance of Self-care Activities (Self-care, 18 items) and takes approximately 15 min to complete.
  Two dimensions of Family Rec are rated on a 5-point Likert scale: frequency of participation (5¼very often to 1¼never) and enjoyment of participation (5¼a great deal to 1¼not at all). ,
  Performance of Self-care Activities are rated on a 5-point Likert scale.
  On the scale , higher scores mean a better outcome.
  For the test-retest reliability, a sub-sample of parents of children with cerebral palsy will complete the measure again two weeks later.

SECONDARY OUTCOMES:
Gross Motor Function Classification System | baseline
  The Gross Motor Function Classification System is a 5-level classification system that describes the gross motor function of children and youth with cerebral palsy on the basis of their self-initiated movement with particular emphasis on sitting, walking, and wheeled mobility. Distinctions between levels are based on functional abilities, the need for assistive technology, including hand-held mobility devices (walkers, crutches, or canes) or wheeled mobility, and to a much lesser extent, quality of movement.
  On the scale , the minimum value is 1 and maximum value 5 and the higher the level the poorer the functional ability of the child.
Manual Ability Classification System | baseline
  The Manual Ability Classification System (MACS) describes how children with cerebral palsy use their hands to handle objects in daily activities. MACS describes five levels. The levels are based on the children's self-initiated ability to handle objects and their need for assistance or adaptation to perform manual activities in everyday life.
  On the scale , the minimum value is 1 and maximum value 5 and the higher the level the poorer the functional ability of the child.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Üniversiteler Mahallesi 1604. Cadde No: 9 Çankaya/ANKARA, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiarello LA, Alghamdi MS, McCoy SW, Avery L, Palisano RJ. Child engagement in daily life measure V2: validation of psychometric properties for children with cerebral palsy. Disabil Rehabil. 2023 Nov;45(23):3912-3921. doi: 10.1080/09638288.2022.2140849. Epub 2022 Nov 2. PMID 36322490
- [Background] Chiarello LA, Palisano RJ, McCoy SW, Bartlett DJ, Wood A, Chang HJ, Kang LJ, Avery L. Child Engagement in Daily Life: a measure of participation for young children with cerebral palsy. Disabil Rehabil. 2014;36(21):1804-16. doi: 10.3109/09638288.2014.882417. Epub 2014 Jan 28. PMID 24467674
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Derived] Simsek Ozguner H, Alkan BM, Gokmen D, Aktas S. Cross-cultural adaptation, validation and reliability of the Turkish version of Child engagement in daily life measure V2 for children with cerebral palsy. Disabil Rehabil. 2026 Jan 1:1-16. doi: 10.1080/09638288.2025.2603833. Online ahead of print. PMID 41477705
- See also: The Child Engagement in Daily Life Measure (Version 2) and conversion tables, which provide an explanation and abbreviated information about the features of the updated version, are available at that link — https://www.canchild.ca/en/research-in-practice/current-studies/on-track/on-track-measures